CLINICAL TRIAL: NCT03615053
Title: Personalized Medicine for Canadians With Hemophilia: a Pragmatic Evaluation of the Web-Accessible Population Pharmacokinetics Service- Hemophilia (WAPPS-Hemo) Tailored Dosing.
Brief Title: Personalized Medicine for Canadians With Hemophilia
Acronym: PMCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PMCH Study
Record Dates: First submitted 2018-07-18; First posted 2018-08-03 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: pharmacokinetics; popPK; PK; Hemophilia
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Intervention Model Description: The PMCH study is a Canadian multicentre, open-label, historically-controlled clinical trial to evaluate the effects of implementing WAPPS-Hemo PopPK-based tailoring of hemophilia prophylaxis regimens using the tailoring dosing function of the WAPPS-Hemo system (WAPPS-Hemo clinical calculator). The study has a non-inferiority design for the primary efficacy and safety outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailored Regimen (Other): Implementation of WAPPS-Hemo personalized dosing regimen.
  Interventions: Other: Implementation of WAPPS-Hemo personalized dosing regimen

INTERVENTIONS:
Other: Implementation of WAPPS-Hemo personalized dosing regimen — Twelve months after enrollment in the study, WAPPS-Hemo will be used to calculate each patients individual pharmacokinetic estimate. Once completed, the WAPPS-Hemo clinical calculator will be used to calculate the optimal regimen based on individual needs.

SUMMARY:
Performing an individual pharmacokinetic (PK) estimate is only the first step in implementing tailored prophylaxis, which requires using the PK profile information to design a personalized treatment regimen matching the treatment needs of individual patients. The overarching goal of WAPPS-Hemo is to provide an easy-to-use web application supporting all the steps needed to accomplish tailoring care of individual patients by matching their unique characteristics to the most appropriate treatment regimen, realizing the promise of personalized medicine.

This study will assess the impact of adopting population PK (popPK) based tailored prophylaxis in clinical practice, including proportion of patients eligible for tailoring, and encountered barriers. The impact on patient important outcomes and on societal outcomes, particularly financial impact, vs. current standardized regimens will be measured. It is hypothesized that WAPPS-Hemo, via estimation of precise individual PK profiles and by supporting the simulation of treatment regimens will:

1. improve or maintain patient important outcomes, while reducing wastage of factor concentrates; and
2. establish best practices and effective knowledge translation strategies for the implementation of personalized medicine.

Additionally, a solid base of data will be generated to model the bleeding risk of severe hemophilia A/B patients undergoing tailored prophylaxis which will enable evaluation of a combination of patient and treatment characteristics predictive of individual bleeding risk.

DETAILED DESCRIPTION:
The PMCH study is a Canadian multicentre, open-label, historically-controlled clinical trial to evaluate the effects of implementing WAPPS-Hemo PopPK-based tailoring of hemophilia prophylaxis regimens using the tailoring dosing function of the WAPPS-Hemo system (WAPPS-Hemo clinical calculator).

The study start date at each centre are staggered by 1-3 months in a modified wedge-shaped design, to allow better differentiation of the effect of the intervention from unrelated but concomitant changes in other aspects of care in the Canadian landscape. Outcomes of interest will be measured for one year prior and for one year after the implementation of the WAPPS-Hemo regimen tailoring procedure.

The two main objectives of this study are:

1. Evaluate the applicability and effectiveness of WAPPS-Hemo PopPK-based tailoring of factor concentrate regimens.
2. Generate a solid base of data to model the bleeding risk of severe hemophilia A/B patients on prophylaxis, evaluating the contribution of patient and treatment characteristics to individual bleeding risk to be reduced by the tailored prophylaxis approach.

PMCH will objectively measure the impact of adopting a PopPK based tailoring of hemophilia treatment. The first goal will be minimizing the occurrence of bleeding events in the hemophilia population. The bleeding rate of Canadian hemophilia patients is still measurable at 2-4 spontaneous joint bleeds per year, which in turn reduce quality of life and consume health resources. It is expected that optimizing treatment goal and modalities will reduce this burden, or at least will not increase it, allowing the pursuit the second goal: minimize the use of resources and prompt a more equitable distribution of factor concentrates. For some patients, standard prophylaxis dosing leads to excessive use of concentrates. It is expected that a small but sizeable proportion of the patient population will be able to successfully reduce their factor concentrate consumption. The third goal will be to generate an evidence-based approach to identify the appropriate target goal(s) for individual patients by modelling the components of their risk of bleeding. Adopting a variable target threshold may enhance objective one and two, maximizing benefits with appropriate allocation of resources.

In addition to WAPPS-Hemo, the study will involve two other tools available to hemophilia treaters in Canada: the Canadian Bleeding Disorders Registry (CBDR) and Patient Reported Outcomes, Burdens and Experiences (PROBE) questionnaire. In particular, this study will leverage the integration of the three tools described above: WAPPS-Hemo, with its ability to generate PK estimates and use them to optimize treatment regiments; CBDR, already collecting most of the information needed to both generate and estimate optimal regimen recommendations for tailoring an individual regimen to meet specified treatment goals; and PROBE, to measure the impact on patient critical life experiences and outcome.

ELIGIBILITY:
Inclusion Criteria:

* individuals with severe congenital hemophilia A and B;
* on continuous factor prophylaxis;
* must be registered on CBDR (iCHIP in BC)

Exclusion Criteria:

* a history of explicit and documented previous treatment tailoring based on pharmacokinetic profiling;
* another congenital or acquired bleeding disorders other than Hemophilia A or B;
* active inhibitors (> 5 Bethesda units) or currently undergoing immune tolerance induction.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in patient quality of life | Completed every 3-6 months for duration of the study, from enrollment to study completion.
  Patient Reported Outcomes, Burdens and Experiences (PROBE) questionnaire. Scores range from 0-1, with a higher value indicating better health status.
Annualized Bleeding Rate (ABR) pre and post-tailoring implementation | Recorded throughout the 2 year duration of the study as they occur.
  ABR from the one year prior to WAPPS-Hemo tailoring to the one-year post-tailoring (absolute number of bleeds per year).

SECONDARY OUTCOMES:
Change in physical activity | Completed every 3-6 months for duration of the study, from enrollment to study completion.
  Patient Reported Outcomes, Burdens and Experiences (PROBE) questionnaire. Scores range from 0-1, with a higher value indicating better health status.
Adherence to prescribed regimen | Recorded throughout the 2 year duration of the study - frequency is as input by patient.
  Measured by comparing the usage resulting from the prescribed regimen, the amount ordered for and dispensed to the patient and the amount logged on the treatment and bleeding diary.
Consumption of factor concentrates | Recorded throughout the 2 year duration of the study - frequency as input by patient.
  Measured as change from the amount prescribed and used before and after the adoption of tailoring.
Feasibility and acceptability of the WAPPS-Hemo based prophylaxis tailoring | Recorded after 1 year at the time of tailoring implementation.
  Measured by proportion of cases with changes in prescribed regimens matching WAPPS-Hemo suggested regimens.
Characteristics of reported bleeds | Recorded throughout the 2 year duration of the study- frequency as input by patient.
  Assessed by exploring information including distribution and typology of joint bleeds as reported in the patient bleed and treatment logs.
Assessment of the predictive performance of the WAPPS-Hemo clinical calculator | Measured within routine clinical practice for 12 months post-tailoring implementation.
  Measured by the comparison of predicted and observed post-infusion levels, when measured as part of routine clinical practice during the study period
Change in joint function | Measured at study enrollment and at 2 years at study completion.
  Measured by the Hemophilia Joint Health Score (HJHS). Scores range from 0-124, with higher values indicating poorer joint health.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Iorio, MD, PhD, FRCPC, Principal Investigator — McMaster University
Locations (6):
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
  - Queen's University, Kingston, Ontario